CLINICAL TRIAL: NCT03927313
Title: Phase IIA Trial of the Safety and Tolerability of Increased Dose Rifampicin and Adjunctive Linezolid With or Without Aspirin, for HIV-associated Tuberculous Meningitis
Brief Title: Linezolid, Aspirin and Enhanced Dose Rifampicin in HIV-TBM
Acronym: LASER-TBM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Robert J Wilkinson, National Principal Investigator, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LASER-TBM
Record Dates: First submitted 2019-03-26; First posted 2019-04-25 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Tuberculosis Meningitis; HIV-1-infection
Keywords: TB meningitis, HIV
MeSH Terms: conditions — Tuberculosis, Meningeal | interventions — Linezolid; Rifampin; Aspirin; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Phase IIA, randomized, active-controlled, open label, parallel-group trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of care anti-tubercular therapy (Active Comparator): Standard of care anti-TB treatment. (10 mg/kg oral rifampicin, 5 mg/kg oral isoniazid, 15 mg/kg oral ethambutol and 25 mg/kg oral pyrazinamide daily for 2 months as fixed dose combination tablets (followed by 10 mg/kg oral rifampicin and 5 mg/kg isoniazid daily for 4-7 months in routine care after study completed)).
  Interventions: Drug: Standard of Care anti-tuberculous therapy; Drug: Dexamethasone
- Intensified anti-tubercular therapy (Experimental): Standard of care anti-TB therapy as described in Arm 1,
  Plus additional 25 mg/kg rifampicin (total dose rifampicin 35 mg/kg orally for the first 56 days of treatment) and linezolid ( 1,200 mg orally daily for first 28 days reduced to 600 mg daily for next 28 days).
  Interventions: Drug: Linezolid; Drug: High dose rifampicin; Drug: Standard of Care anti-tuberculous therapy; Drug: Dexamethasone
- Intensified anti-tubercular therapy plus aspirin (Experimental): Standard of care anti-TB therapy as described in Arm 1,
  Plus additional 25 mg/kg rifampicin (total dose rifampicin 35 mg/kg orally for the first 56 days of treatment) and linezolid ( 1,200 mg orally daily for first 28 days reduced to 600 mg daily for next 28 days),
  Plus aspirin (1000mg orally daily for the first 56 days of Tuberculous Meningitis treatment)
  Interventions: Drug: Linezolid; Drug: High dose rifampicin; Drug: Aspirin; Drug: Standard of Care anti-tuberculous therapy; Drug: Dexamethasone

INTERVENTIONS:
Drug: Linezolid — For both experimental arms: 1.2g linezolid 28 days, followed by 600mg linezolid for 28 days
  Arms: Intensified anti-tubercular therapy; Intensified anti-tubercular therapy plus aspirin
Drug: High dose rifampicin — For both experimental arms: additional 25mg/kg (making a total of 35mg/kg) rifampicin, for the first 56 days of treatment
  Arms: Intensified anti-tubercular therapy; Intensified anti-tubercular therapy plus aspirin
Drug: Aspirin — For only one of the experimental arms: 1000mg of aspirin daily for 56 days.
  Arms: Intensified anti-tubercular therapy plus aspirin
Drug: Standard of Care anti-tuberculous therapy — 10mg/kg oral rifampicin, 5mg/kg oral isoniazid, 15mg/kg oral ethambutol, 25mg/kg oral pyrazinamide daily for 56 days.
Drug: Dexamethasone — Dexamethasone according to doses of Thwaites criteria for the first 8 weeks of anti-tuberculous treatment. Doses differ according to participants Medical Research Council (MRC) grade. Given orally if participant can swallow and intravenously if they cannot.

SUMMARY:
LASER-TBM is a parallel group, randomized, multi-arm phase IIa trial evaluating the safety of increased dose rifampicin (RIF) plus linezolid (LZD), with or without aspirin (ASA), for the treatment of HIV-infected adults with tuberculous meningitis (TBM). The study will recruit 100 HIV-infected adults with TBM across four sites in South Africa.

The primary endpoint is the occurrence of solicited treatment-related adverse events.

Secondary endpoints include death and disability (including neurocognitive impairment), radiological outcomes, and the occurrence of immune reconstitution inflammatory syndrome (IRIS).

A nested pharmacokinetic (PK) substudy aims to:

1. Describe the plasma and cerebrospinal fluid (CSF) PK of LZD and high dose RIF.
2. Evaluate the relationship between drug exposures, toxicity and efficacy.
3. Compare exposures between intravenous and oral RIF administration.
4. Investigate the impact of high dose RIF on LZD and dolutegravir (DTG).

DETAILED DESCRIPTION:
HIV-1 infected adults with newly-diagnosed TBM (n = 100) will be recruited from four public-sector hospitals in Cape Town and Port Elizebeth, South Africa. Participants will be randomised across two experimental (n = 30 each) and one standard of care (n = 40) arms. Treatment will be provided in all arms for 56 days, after which participants will be referred back to public sector facilities to complete standard therapy for HIV-associated TBM.

The primary objective of the study is to investigate the safety of enhanced antimicrobial therapy including increased dose RIF and LZD with or without adjunctive aspirin added to standard therapy for TBM in HIV-1 infected adults.

Secondary objectives are;

1. To determine cerebrospinal fluid M.tb culture positivity and Gene Xpert® Ultra positivity at baseline and at 3 and 28 days post treatment by allocation.
2. To evaluate the effect of aspirin and enhanced tuberculosis treatment on the incidence of immune reconstitution syndrome in participants starting antiretroviral therapy.
3. To evaluate the effect of high dose rifampicin and linezolid, with and without aspirin on the transcriptional signature derived from whole blood and cerebrospinal fluid RNA sequencing, as well as the metabolomic and proteomic profiles, in tuberculous meningitis.
4. To evaluate the effect of high dose rifampicin and linezolid with and without aspirin on central nervous system imaging in conjunction with clinical, immunological and transcriptional profiling.
5. To store biological samples for future analysis of potential biomarkers of treatment efficacy and/or novel diagnostic assays.
6. To determine i) whether host genotype, including LTA4H genotype, influences therapeutic effect of aspirin in HIV-TBM and ii) the pharmacogenetic influence on rifampicin and linezolid exposures and toxicity.

All participants will receive antitubercular chemotherapy and corticosteroids as standard of care as per national South African guidelines. Participants allocated to experimental arms 2 and 3 will receive additional rifampicin (total oral dose 35 mg/kg/day) plus oral linezolid 1200mg daily for the first 28 days, reduced to 600 mg daily for the next 28 days. Those randomized to experimental arm 3 will also receive oral aspirin 1000 mg daily.

All consenting LASER-TBM participants in experimental arms (n = 60) will undergo a second randomisation to receive either oral (35mg/kg) or IV (20mg/kg) rifampicin at the time of study entry. This sub-study is powered to demonstrate bioequivalence at day 3 of administration, after which all participants will be continued on oral rifampicin dosed at 35mg/kg.

Trial participation will be for 180 days post-randomization: primary safety endpoints and secondary efficacy endpoints will be evaluated at day 56; additional secondary endpoints will be evaluated at day 180.

There are seven scheduled study visits. The first six of thee will occur within the first 56 days, with an additional structured interview at 6 months. All visits will involve a clinical assessment including specified clinical outcome measures to assess functional and cognitive disability. Phlebotomy will be performed at study visits within the first 56 days to monitor for pre-specified parameters of drug safety (haematology, biochemistry) as well as to collect blood for downstream transcriptomic, proteomic and metabolomic analysis. Lumbar puncture will take place at day 3 and day 28. Cerebrospinal fluid will be analysed for Mycobacterium tuberculosis culture and Gene Xpert® Ultra cycle threshold values. Cerebrospinal fluid (CSF) will be stored for downstream transcriptomic, proteomic and metabolomic analysis. Baseline and day 56 brain imaging will be performed in all study participants.

All enrolled participants will undergo sparse plasma PK sampling at the Day 28 and Day 56 visits.

Cerebrospinal fluid (CSF) will be collected from all participants for determination of linezolid and rifampicin concentrations on Days 3 and 28. The timing of the Day 3 lumbar puncture will be randomised to intervals of 1 - 3, 3 - 6, 6 - 10, and 24 hours after observed antitubercular drug dosing in order to construct a concentration-time profile for the population. A single sample will be collected at each time interval. A second lumbar puncture will take place at the Day 28 visit, to coincide with the 4-hour plasma PK sample.

All participants (n=100) will be offered participation in the intensive sampling component of the PK sub-study at the time of randomization to the main study. Intensive plasma sampling will take place at the Day 3 study visit. Serial venous blood samples will be collected through a peripheral intravenous catheter pre-dose, and at 0.5, 1, 2, 3, 6, 8 - 10, and 24 hours after witnessed drug intake and an overnight fast. Sparse sampling will be performed at Day 3 for participants who decline intensive sampling or in whom this fails.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 seropositivity by rapid test, confirmed by enzyme-linked immunosorbent assay (regardless of Antiretroviral Therapy (ART) status);
* Age 18 years or older;
* Tuberculous meningitis defined as 'possible', 'probable' or 'definite' as per published case definitions

Exclusion Criteria:

* Rifampicin-resistant M. tb detected in any microbiological specimen;
* History of allergy or hypersensitivity to H, E, R and Z, LZD or ASA;
* Received more than 5 days of antitubercular therapy in the 30 days prior to screening;
* Received a dose of ASA or any other NSAID within 2 weeks of screening;
* CSF unobtainable by lumbar puncture or another procedure;
* Evidence of bacterial or cryptococcal meningitis;
* Severe concurrent uncontrolled opportunistic infection including but not limited to active cytomegalovirus-associated disease, Kaposi sarcoma, Pneumocystis jirovecii pneumonia, HIV related or unrelated malignancy or gastrointestinal bleeding;
* Any other form of immunosuppressive therapy including antineoplastic and biologic agents apart from corticosteroids;
* Is pregnant in the third trimester;
* Peripheral neuropathy scoring Grade 3 or above on Brief Peripheral Neuropathy Score
* Any disease or condition in which the use of the standard TB drugs or any of their components is contraindicated, including but not limited to allergy to any TB drug or their components;
* The presence of one or more of the following:

  * Estimated glomerular filtration rate (eGFR) < 20ml/min/1.73m2 (using the Cockcroft-Gault equation)
  * International normalised ration (INR) > 1.4 and/or clinical evidence of liver failure or decompensated cirrhosis
  * Hemoglobin < 8.0 g/dL
  * Platelets < 50 x109 /L
  * Neutrophils < 0.5 x 109 cells/L;
* The patient has any disease or condition in which any of the medicinal products listed in the section pertaining to prohibited medication is used and cannot be safely stopped;
* The patient has a known or suspected, current or history of drug abuse, within the past 2 years, that is, in the opinion of the investigators, sufficient to compromise the safety or cooperation of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants in each arm who develop treatment related adverse events (AEs). | 56 days
  The amount of participants who develop any of the following treatment related adverse events by the time they have been on treatment for 56 days will be counted: Peripheral neuropathy, optic neuropathy, anaemia, neutropaenia, thrombocytopaenia, upper gastro-intestinal haemorrhage, intracerebral haemorrhage, drug-induced liver injury.

SECONDARY OUTCOMES:
Death and disability after 56 days on treatment. | 56 days
  A comparison will be made of the proportion of participants in each arm who died, and their grade of disability will be compared according to Modified Rankin Scoring.
Death at day 56 and day 180. | 180 days
  In all arms: the number of participants who have died at Day 56 will be compared to those that have died at Day 180.
Number of participants who are disabled. | 180 days
  Comparison of level of disability of participants at 56 and 180 days, stratifying by Medical Research Council grade.
Number of participants who develop Grade 3 or Grade 4 adverse events (AEs). | 56 days
  In all 3 arms: comparison of the number of participants who develop Grade 3 or Grade 4 adverse events (according to Division of AIDS (DAIDS) criteria) by the time they have been on treatment or 56 days.
Number of participants in whom experimental drugs had to be stopped. | 56 days
  At 56 days on treatment, the number of participants in the experimental arms in whom rifampicin, linezolid and/or aspirin had to be stopped.
Linezolid toxicity | 56 days
  To note the presence of the following adverse events in all participants in the experimental arms: peripheral neuropathy, optic neuropathy, anaemia, neutropaenia, thrombocytopaenia and hyperlactataemia.
Major bleeding events. | 180 days
  To note at 6 months, the amount of participants who develop upper gastro-intestinal or intra-cerebral haemorrhage after receiving 1000mg daily aspirin as part of the trial.
Cerebrospinal fluid culture conversion. | Day 28 and day 56
  To compare in the different arms, between lumbar punctures done at day 3 and day 28, the time to automated liquid culture positivity and Gene-Xpert ultra threshold values (for mycobacterium tuberculosis) of cerebrospinal fluid.
The occurrence of TBM-immune reconstitution inflammatory syndrome | 56 days
  The amount of participants in all 3 arms who develop paradoxical tuberculosis immune reconstitution, as defined by th modified INSHI criteria.
Changes on brain imaging | Day 56
  To compare at day 56, in participants who had brain imaging at baseline, changes in brain imaging at day 56.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Wilkinson, PhD, Principal Investigator — Wellcome Centre for Infectious Diseases Research in Africa, Institute of Infectious Disease and Molecular Medicine, University of Cape Town; Sean Wasserman, MMed, Principal Investigator — Wellcome Centre for Infectious Diseases Research in Africa, Institute of Infectious Disease and Molecular Medicine, University of Cape Town; Graeme Meintjes, PhD, Principal Investigator — Wellcome Centre for Infectious Diseases Research in Africa, Institute of Infectious Disease and Molecular Medicine, University of Cape Town; John Black, MBChB, Principal Investigator — Department of Medicine, University of Cape Town and Walter Sisal University; Angharad G Davis, Dr, Study Chair — 1. Faculty of Life Sciences, University College London, UK 2. Department of Medicine, University of Cape Town, Observatory 7925, Republic of South Africa
Locations (4):
- South Africa (4):
  - Livingstone Hospital, Port Elizabeth, Eastern Cape
  - Mitchells Plain Hospital, Cape Town, Western Cape
  - Groote Schuur Hospital, Cape Town, Western Cape
  - New Somerset Hospital, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Abdelgawad N, Wasserman S, Abdelwahab MT, Davis A, Stek C, Wiesner L, Black J, Meintjes G, Wilkinson RJ, Denti P. Linezolid Population Pharmacokinetic Model in Plasma and Cerebrospinal Fluid Among Patients With Tuberculosis Meningitis. J Infect Dis. 2024 Apr 12;229(4):1200-1208. doi: 10.1093/infdis/jiad413. PMID 37740554
- [Derived] Davis AG, Wasserman S, Stek C, Maxebengula M, Jason Liang C, Stegmann S, Koekemoer S, Jackson A, Kadernani Y, Bremer M, Daroowala R, Aziz S, Goliath R, Lai Sai L, Sihoyiya T, Denti P, Lai RPJ, Crede T, Naude J, Szymanski P, Vallie Y, Banderker IA, Moosa MS, Raubenheimer P, Candy S, Offiah C, Wahl G, Vorster I, Maartens G, Black J, Meintjes G, Wilkinson RJ. A Phase 2A Trial of the Safety and Tolerability of Increased Dose Rifampicin and Adjunctive Linezolid, With or Without Aspirin, for Human Immunodeficiency Virus-Associated Tuberculous Meningitis: The LASER-TBM Trial. Clin Infect Dis. 2023 Apr 17;76(8):1412-1422. doi: 10.1093/cid/ciac932. PMID 36482216
- [Derived] Davis AG, Wasserman S, Maxebengula M, Stek C, Bremer M, Daroowala R, Aziz S, Goliath R, Stegmann S, Koekemoer S, Jackson A, Lai Sai L, Kadernani Y, Sihoyiya T, Liang CJ, Dodd L, Denti P, Crede T, Naude J, Szymanski P, Vallie Y, Banderker I, Moosa S, Raubenheimer P, Lai RPJ, Joska J, Nightingale S, Dreyer A, Wahl G, Offiah C, Vorster I, Candy S, Robertson F, Meintjes E, Maartens G, Black J, Meintjes G, Wilkinson RJ. Study protocol for a phase 2A trial of the safety and tolerability of increased dose rifampicin and adjunctive linezolid, with or without aspirin, for HIV-associated tuberculous meningitis [LASER-TBM]. Wellcome Open Res. 2021 Jun 1;6:136. doi: 10.12688/wellcomeopenres.16783.1. eCollection 2021. PMID 34286103
- [Derived] Wasserman S, Davis A, Stek C, Chirehwa M, Botha S, Daroowala R, Bremer M, Maxebengula M, Koekemoer S, Goliath R, Jackson A, Crede T, Naude J, Szymanski P, Vallie Y, Moosa MS, Wiesner L, Black J, Meintjes G, Maartens G, Wilkinson RJ. Plasma Pharmacokinetics of High-Dose Oral versus Intravenous Rifampicin in Patients with Tuberculous Meningitis: a Randomized Controlled Trial. Antimicrob Agents Chemother. 2021 Jul 16;65(8):e0014021. doi: 10.1128/AAC.00140-21. Epub 2021 Jul 16. PMID 33972248